CLINICAL TRIAL: NCT06586879
Title: Psychiatric Comorbidities in Children and Adolescent Patients with Diabetes Mellitus Type 1.
Brief Title: Psychiatric Comorbidities in Type 1 Diabetes Mellitus.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omnia Mohamed Fath-Allah, Resident doctor, Assiut University
Other Study IDs: Psychiatry in type 1 DM
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
This study aimed to assess the prevalence of psychiatric comorbidities in children and adolescents with diabetes mellitus type 1.

Assessing the impact of diabetes mellitus type 1 on quality of life. And determine the effect of associated factors on the development of psychiatric comorbidities and on quality of life in diabetes mellitus type 1.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (TDM) is a chronic autoimmune disease. that affected carbohydrate metabolism and caused by insulin insufficiency resulting in increased blood glucose. It's one of the most common endocrine and metabolic conditions in childhood. There's 9 million people live with T1DM worldwide according to International Diabetes Federation. In Egypt, 1 in 98 families are impacted and the disease is growing at 6.7% each year. Living with T1DM has been associated with a significant impact on a person's social, mental, and psychological quality of life (QoL). as the individual must adopt blood glucose monitoring, use of injections or diabetes technology for insulin regulation, diet restrictions, and exercise. Also, there's increased risk of developing micro-and macro-vascular complications that result in morbidity and mortality in Long-term uncontrolled DM. therefore, these children and adolescents with T1DM have an increased risk of psychiatric comorbidities like depression, anxiety and sleep disorders, depression is one of the most common disorders. They appear to have a greater incidence of depression, anxiety and poor health-related quality of life (HRQoL) compared to their healthy peers. This is associated with suboptimal diabetes outcomes and better metabolic control has been found to correlate with better quality of life. This occurs especially when diagnosed at earlier age of onset, history of severe hypoglycemia and chronic hyperglycemia. There are no available studies that assess the presence of psychiatric comorbidities in T1DM in our locality.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged between 8 and 15 years, diagnosed with diabetes mellitus type 1 and on medical treatment.

Exclusion Criteria:

* Patients with major psychiatric disorders or have cognitive difficulties.
* Patients unable or refuse to give consent.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescent Patients with type 1 diabetes medllitus aged 8-15 years old.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The prevalence of psychiatric comorbidities in children and adolescents with diabetes mellitus type 1. | 2 years
  This outcome will be measured using:
  The Kiddie-Schedule for Aﬀective Disorders and Schizophrenia for School-Age Children-Present and Lifetime (K-SADS-PL) version
the prevalence of depression, anxiety and sleep disorder in children and adolescents with diabetes mellitus type 1 | 2 years
  this outcome will be measured using:
  1. Children's Depression Inventory 2 Self Report-Short (CDI-2) (12)
  2. The Spence Children's Anxiety Scale
  3. Children's Sleep Habits Questionnaire (CSHQ)

SECONDARY OUTCOMES:
The impact of diabetes mellitus type 1 on quality of life. | 2 years
  This outcome will be measured using:
  Pediatric quality of life inventory 4.0 genetic Core scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Mahran, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashraf MN, Cheng AYY, Robinson DJ. Emotional, Psychological, and Social Well-being Experience of Long-Term Living with Type 1 Diabetes Mellitus: A Patient-Psychiatrist-Endocrinologist Perspective. Diabetes Ther. 2024 Feb;15(2):317-323. doi: 10.1007/s13300-023-01527-w. Epub 2024 Jan 17. PMID 38233629
- [Background] Abouzid MR, Ali K, Elkhawas I, Elshafei SM. An Overview of Diabetes Mellitus in Egypt and the Significance of Integrating Preventive Cardiology in Diabetes Management. Cureus. 2022 Jul 20;14(7):e27066. doi: 10.7759/cureus.27066. eCollection 2022 Jul. PMID 36000101
- [Background] El-Ziny MA, Salem NA, El-Hawary AK, Chalaby NM, Elsharkawy AA. Epidemiology of childhood type 1 diabetes mellitus in Nile Delta, northern Egypt - a retrospective study. J Clin Res Pediatr Endocrinol. 2014;6(1):9-15. doi: 10.4274/Jcrpe.1171. PMID 24637304
- See also: Type 1 diabetes in international diabetes Federation — https://idf.org/about-diabetes/type-1-diabetes/
- See also: Type 1 diabetes index — https://www.t1dindex.org/countries/egypt/
- See also: Psychological care of children and adolescents with type 1 diabetes — https://pubmed.ncbi.nlm.nih.gov/30058247/
- See also: Evaluation of psychological characteristics of Turkish children with type 1 diabetes mellitus from two demographically and geographically distinct regions — https://pubmed.ncbi.nlm.nih.gov/30968638/
- See also: The cognitive and psychological effects of living with type 1 diabetes — https://pubmed.ncbi.nlm.nih.gov/31850538/
- See also: High Rate of Depression among Saudi Children with Type 1 Diabetes — https://pubmed.ncbi.nlm.nih.gov/34770232/
- See also: Updating and validation of the socioeconomic status scale for health research in Egypt — https://pubmed.ncbi.nlm.nih.gov/23057390/
- See also: Type 1 Diabetes — https://www.ncbi.nlm.nih.gov/books/NBK507713/
- See also: Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data — https://pubmed.ncbi.nlm.nih.gov/9204677/
- See also: Children's Depression Inventory 2nd Edition — https://www.apa.org/obesity-guideline/depression-inventory.pdf
- See also: A measure of anxiety symptoms among children — https://pubmed.ncbi.nlm.nih.gov/9648330/
- See also: CHILDREN'S SLEEP HABITS QUESTIONNAIRE (ABBREVIATED) — https://njaap.org/wp-content/uploads/2016/04/Childrens-Sleep-Habits-Questionnaire.pdf
- See also: The PedsQL 4.0 Generic Core Scales: — https://pubmed.ncbi.nlm.nih.gov/11977437/